CLINICAL TRIAL: NCT05340231
Title: An Exploratory Study of Sequential Transarterial Chemoembolization With Lipiodol and Neoadjuvant Chemotherapy in the Treatment of Initial Unresectable Colorectal Cancer
Brief Title: An Exploratory Study of Sequential Transarterial Chemoembolization With Lipiodol and Neoadjuvant Chemotherapy in the Treatment of Initial Unresectable Colorectal Cancer (CRC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gang Wu (Other)
Responsible Party: Sponsor-Investigator, Gang Wu, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC-2022-01
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): sequential transarterial chemoembolization with lipiodol and neoadjuvant chemotherapy
  Interventions: Drug: TACE protocol
- Control group (Active Comparator): neoadjuvant chemotherapy alone
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: TACE protocol — Transarterial infusion chemotherapy: Oxaliplatin(85mg/m^2)+Raltitrexed(3mg) Chemoembolization: Lipiodol emulsion (lipiodol 10ml+ Oxaliplatin 85mg +Lidocaine 1ml)，The endpoint for embolization was defined as stagnation of blood flow of the posterior mesenteric artery.
  Intervention cycle：4W; Treatment times: 2. followed by mFOLFOX6
  Arms: Study group
Drug: Neoadjuvant Chemotherapy — mFOLFOX6, Q2W
  Arms: Control group

SUMMARY:
This is a prospective, open-labelled study to evaluate the efficacy and safety of sequetial transarterial chemoembolization with lipiodol and neoadjuvant chemotherapy in the treatment of initial unresectable colorectal cancer. The progression-free-survival (PFS) will be evaluated as the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Has fully understood and voluntarily signed an written Informed Consent and agreed to follow the research plan treatment and visiting plan;
2. Aged >=18 years, <= 85 years;
3. Histologically confirmed initial unresectable colorectal cancer;
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
5. Expected survival period ≥ 3 months;
6. At least one measurable lesion, according to RECIST 1.1;
7. The main function is normal.

Exclusion Criteria:

1. Known hypersensitivity to any of the study drugs or excipients;
2. Hypertension that is not controlled by the drug;
3. International normalized ratio (INR) > 1.5 or partially activated prothrombin time (APTT) > 1.5 × ULN;
4. WBC count < 3000 /mm^3;
5. Platlet count < 50000 /mm^3;
6. Poorly controlled diabetes before enrollment;
7. Clinically significant electrolyte abnormalities judged by researchers;
8. Patients with obvious evidence of bleeding tendency or medical history of hematochezia within 3 months before enrollment;
9. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%;
10. Active infection or serious infection that is not controlled by drug;
11. History of clinically significant hepatic disease (ALT and/or AST >5 times the upper normal limit);
12. Women who are pregnant or lactating;
13. Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0g;
14. Have any other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other conditions, which according to the judgment of the investigator, it is reasonable to suspect that the patient is not suitable for the use of the study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
ORR | up to 3 years
  ORR is defined as the percentages of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria
Overall survival (OS) | up to 3 years
  The time from recruitment to death due to any cause.
Pathological response rate (PCR+MPR) | up to 3 years
  Pathologic complete response (pCR) was defined as absence of viable tumor in the post-treatment surgical specimens and major pathologic response (MPR) was defined as ≤ 10% viable tumor.

IPD SHARING:
Plan to Share IPD: No